CLINICAL TRIAL: NCT02120872
Title: Platelet - Rich Fibrin Combined With 1.2mg Simvastatin for the Treatment of 3 - Wall Intrabony Defects in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin Combined With Simvastatin for Treatment of Intrabony Defect in Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head of Department, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2011-2012/E
Record Dates: First submitted 2014-04-17; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Three Wall Intrabony Defects in Chronic Periodontitis
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRF and SMV Group (Active Comparator): sites treated with Open Flap Debridement with Platelet Rich Fibrin along with Simvastatin
  Interventions: Drug: Platelet rich fibrin and simvastatin
- PRF Group (Sham Comparator): sites treated with Open Flap Debridement with autologous Platelet Rich Fibrin
  Interventions: Biological: Platelet rich fibrin
- OFD Group (Other): sites treated with Open Flap Debridement i.e. conventional flap surgery
  Interventions: Procedure: Open Flap Debridement alone

INTERVENTIONS:
Drug: Platelet rich fibrin and simvastatin — Three wall intrabony defect sites treated with Open Flap Debridement. 0.1 mL prepared SMV gel (1.2 mg/0.1 mL) was mixed with PRF. The PRF - SMV mixture was delivered to the defect.
  Arms: PRF and SMV Group
Biological: Platelet rich fibrin — Three wall intrabony defect sites treated with Open Flap Debridement. PRF was placed into the intrabony defect.
  Arms: PRF Group
Procedure: Open Flap Debridement alone — Three wall intrabony defect sites treated with Open Flap Debridement only. No PRF or SMV was delivered to the defect.
  Arms: OFD Group

SUMMARY:
The purpose of the present study was to investigate the efficacy of autologous Platelet rich fibrin (PRF) or PRF and Simvastatin (SMV) with open flap debridement (OFD) in the treatment of three wall intrabony defects in comparison to OFD alone.

DETAILED DESCRIPTION:
90 systemically healthy subjects were divided randomly into three groups (30 subjects in each group, per subject one site). Control group consisted of the sites treated with OFD and test groups sites were treated with OFD with autologous PRF or PRF with SMV. Site-specific plaque index (PI), sulcus bleeding index (mSBI), probing depth (PD), relative attachment level (RAL) and intrabony defect (IBD) depth reduction was measured at baseline and 9 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the diagnosis of chronic periodontitis
* presence of three walled intrabony defects (IBD) ≥ 3 mm deep (distance between alveolar crest and base of the defect on intraoral periapical radiograph [IOPA])
* interproximal probing depth (PD) ≥ 5 mm following scaling and root planing (SRP) in asymptomatic tooth

Exclusion Criteria:

* Subjects, with the diagnosis of aggressive periodontitis,
* with known systemic illness and taking medications known to affect the outcomes of periodontal therapy
* insufficient platelet count (< 200,000/mm3),
* pregnancy / lactation
* use of any form of tobacco
* unacceptable oral hygiene (if plaque index [PI] (Silness & Loe 1964) >1.5) after the reevaluation of phase I therapy
* teeth with furcation defects
* non-vital
* mobility of tooth ≥ Grade II

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study was defect depth reduction evaluated radiographically | At baseline and 9 month after surgery

SECONDARY OUTCOMES:
Probing Depth | At baseline and 9 month after surgery
Relative Attachment Level | At baseline and 9 month after syrgery
modified Sulcul Bleeding Index | At baseline and 9 month after surgery
Plaque Index | At baseline and 9 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — Government Dental College and Research Institute, Bangalore
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India